CLINICAL TRIAL: NCT04741776
Title: A Pilot Randomized Trial of Video-based Family Therapy for Home Visited Mothers With Perinatal Depressive Symptoms
Brief Title: A Pilot Randomized Trial of Video-based Family Therapy for Depressed Home Visited Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Fallon P. Cluxton-Keller, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D21065; 1R34MH124951 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Perinatal Depression; Postpartum Depression; Family Conflict
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based family therapy (Experimental): Resilience Enhancement Skills Training (REST)
  Interventions: Behavioral: Resilience Enhancement Skills Training
- Standard of care (Active Comparator): Video-based Problem Solving individual Therapy (V-PST)
  Interventions: Behavioral: Problem-Solving Individual Therapy

INTERVENTIONS:
Behavioral: Resilience Enhancement Skills Training — Family therapy
  Arms: Video-based family therapy
Behavioral: Problem-Solving Individual Therapy — Individual therapy
  Arms: Standard of care

SUMMARY:
Depressed mothers (pregnant and post-delivery) make up a significant portion of Maternal, Infant, and Early Childhood Home Visiting (MIECHV) clients. Home visited mothers often experience family conflict that precipitates or worsens their depressive symptoms. This study uses an effectiveness-implementation hybrid type 1 design with a pilot randomized trial to test the feasibility, acceptability, tolerability, safety, and preliminary effectiveness of an innovative family therapy intervention that uses technology to bypass barriers to increase access to treatment for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Mothers in any trimester of pregnancy through 18 months postpartum who are enrolled in home visiting at a participating agency;
* Fluent in English;
* Mother and her family member have at least an 8th grade education;
* Mothers with Beck Depression Inventory-Second Edition scores of at least 20;
* Perceived Hostility Survey-Adult raw scores of at least 16 for the adult mother and her adult family member; Perceived Hostility Survey-Child raw scores of at least 14 for the adolescent mother and her adolescent intimate partner; and
* Consistent internet access on their cell phones, tablets, or computer equipped with a microphone and camera.

Exclusion Criteria:

* Suicidal ideation in the mother and/or her family member;
* Mothers with bipolar disorder symptoms;
* Psychotic symptoms in the mother and/or her family member;
* Mother is currently receiving individual therapy;
* Family is currently receiving family therapy;
* Mothers who have been taking an antidepressant for less than 2 months; and
* Families with domestic violence.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fallon Cluxton-Keller, Ph.D., Principal Investigator — Dartmouth-Hitchcock Clinic
Locations (1):
- Dartmouth-Hitchcock Clinic, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Cluxton-Keller F, Xie H, Hegel MT, Donnelly CL, Bruce ML. Preliminary Effectiveness of Family Therapy for Perinatal Depressive Symptoms: Results From a Pilot Randomized Trial. Fam Process. 2025 Jun;64(2):e70032. doi: 10.1111/famp.70032. PMID 40159324
- [Derived] Cluxton-Keller F, Hegel MT, Donnelly CL, Bruce ML. Video-Delivered Family Therapy for Perinatal Women With Depressive Symptoms and Family Conflict: Feasibility, Acceptability, Safety, and Tolerability Results From a Pilot Randomized Trial. JMIR Form Res. 2023 Nov 3;7:e51824. doi: 10.2196/51824. PMID 37921846
- [Derived] Cluxton-Keller F, Hegel MT. A Video-Delivered Family Therapeutic Intervention for Perinatal Women With Clinically Significant Depressive Symptoms and Family Conflict: Indicators of Feasibility and Acceptability. JMIR Form Res. 2022 Oct 4;6(10):e41697. doi: 10.2196/41697. PMID 36194458

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Research staff obtained electronic consent of the IRB-approved consent forms for the eligibility screen and study enrollment from willing participants
Pre-assignment Details: The mother, and her family member, were randomized to one of two study groups: 1) video-based family therapy (Resilience Enhancement Skills Training, REST), or 2) standard of care (Video-based Problem Solving individual Therapy, V-PST). REST is designed for participation by the dyad. By design, only the mother participated in V-PST sessions. The Enrollment number and Started/Completed number represents individual participants.
Groups:
- Video-based Family Therapy: Mothers; Video-based Family Therapy: Family Members: Resilience Enhancement Skills Training (REST) is the family therapy intervention. Mothers and their family members participated in REST sessions. Study measures were administered to each mother and her family member, separately.
- Standard of Care: Mothers; Standard of Care: Family Members: Video-based Problem-Solving individual Therapy (V-PST) is the active comparison condition. Only mothers participated in V-PST sessions. Study measures were administered to each mother and her family member, separately.
Period: Overall Study
Arm/Group | Video-based Family Therapy: Mothers | Video-based Family Therapy: Family Members | Standard of Care: Mothers | Standard of Care: Family Members
Started | 42 | 42 | 41 | 41
Started Assigned Intervention | 38 | 38 | 37 | 37
Completed (contributed 6 month follow-up data) | 35 | 32 | 30 | 24
Not Completed | 7 | 10 | 11 | 17
Not completed — Withdrawal by Subject | 7 | 10 | 10 | 17
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video-based Family Therapy: Mothers | Video-based Family Therapy: Family Members | Standard of Care: Mothers | Standard of Care: Family Members | Total
Number analyzed (Participants) | 42 | 42 | 41 | 41 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1 | 0 | 2
  Between 18 and 65 years | 41 | 41 | 40 | 40 | 162
  >=65 years | 0 | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (5.7) | 33.1 (11.4) | 28.3 (5.5) | 38.0 (14.6) | 31.79 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 5 | 41 | 13 | 101
  Male | 0 | 37 | 0 | 28 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 4 | 7
  Not Hispanic or Latino | 42 | 39 | 41 | 37 | 159
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 2 | 7
  Asian | 2 | 2 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 2 | 1 | 1 | 1 | 5
  White | 28 | 25 | 28 | 25 | 106
  More than one race | 9 | 12 | 7 | 11 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 42 | 41 | 41 | 166

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Depressive Symptoms on the Beck Depression Inventory-Second Edition at Six Month Follow-up
Description: Maternal depressive symptoms. The Beck Depression Inventory-Second Edition scores range from 0 (no depressive symptoms) to 63 (severe depressive symptoms).
  Higher score indicates greater depressive symptoms.
Time Frame: Baseline and six month follow-up
Population: All mothers who attended at least 1 session.
Measure: Mean (Standard Deviation); unit: units on a scale (BDI-II)
Groups:
- Video-based Family Therapy: Mothers: Resilience Enhancement Skills Training (REST) is the family therapy intervention. Mothers and their family members participated in REST sessions.
- Standard of Care: Mothers: Video-based Problem-Solving individual Therapy (V-PST) is the active comparison condition. Only mothers participated in V-PST sessions.
Arm/Group | Video-based Family Therapy: Mothers | Standard of Care: Mothers
Number analyzed (Participants) | 38 | 37
units on a scale (BDI-II)
  Baseline | 28.3 (5.8) | 27.0 (6.1)
  Six Month Follow-Up | 6.9 (4.9) | 13.2 (8.6)

2. Primary Outcome: Change From Baseline in Family Conflict on the Perceived Hostility Survey at the Six Month Follow-up
Description: Family conflict was measured using the Perceived Hostility Survey (Ages 18 +) and Perceived Hostility Survey (Ages 8-17). In both versions of the Perceived Hostility Survey, raw scores are converted to uncorrected T-scores. Scores one standard deviation or more below the mean (T ≤ 40) suggest low levels of perceived hostility and scores one standard deviation or more above the mean (T ≥ 60) suggest high levels of perceived hostility.
Time Frame: baseline and six month follow-up
Measure: Number; unit: T-score
Groups:
- Video-based Family Therapy:Family Members: Resilience Enhancement Skills Training (REST) is the family therapy intervention. Mothers and their family members participated in REST sessions. Study measures were administered to each mother and her family member, separately.
- Standard of Care:Mothers; Standard of Care:Family Members: Video-based Problem-Solving individual Therapy (V-PST) is the active comparison condition. Only mothers participated in V-PST sessions. Study measures were administered to each mother and her family member, separately.
Arm/Group | Video-based Family Therapy: Mothers | Video-based Family Therapy:Family Members | Standard of Care:Mothers | Standard of Care:Family Members
Number analyzed (Participants) | 38 | 38 | 37 | 37
T-score
  Baseline | 58.7 | 60.1 | 60.1 | 58.7
  Six month follow-up | 44.2 | 46.3 | 52.9 | 52.9

3. Primary Outcome: Change From Baseline in Family Cohesion on the Multidimensional Scale of Perceived Social Support-Family at the Six Month Follow-up
Description: Family cohesion was measured using the Multidimensional Scale of Perceived Social Support-Family with scores that range from 7-28. Higher scores indicate greater cohesion.
Time Frame: baseline and six month follow-up
Population: All participants who completed at least one session. By design, mothers' family members did not participate in the Standard of Care intervention sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Video-based Family Therapy:Mothers; Video-based Family Therapy: Family Members: Resilience Enhancement Skills Training (REST) is the family therapy intervention. Mothers and their family members participated in REST sessions. Study measures were administered to each mother and her family member, separately.
Arm/Group | Video-based Family Therapy:Mothers | Video-based Family Therapy: Family Members | Standard of Care:Mothers | Standard of Care:Family Members
Number analyzed (Participants) | 38 | 38 | 37 | 37
units on a scale
  Baseline | 20.6 (3.7) | 20.9 (4.3) | 19.7 (5.1) | 20.2 (4.0)
  Six month follow-up | 23.7 (3.4) | 24.0 (2.8) | 19.3 (6.0) | 20.9 (6.7)

4. Primary Outcome: Change From Baseline in Cognitive Reappraisal on the Emotion Regulation Questionnaire-Cognitive Reappraisal Scale at Six Month Follow-up
Description: Family cognitive reappraisal. Adult participants completed the Emotion Regulation Questionnaire-Cognitive Reappraisal scale (Adult version) with scores that range from 6 (infrequent use of cognitive reappraisal) to 42 (frequent use of cognitive reappraisal). Adolescent participants completed the Emotion Regulation Questionnaire-Cognitive Reappraisal scale (Children and Adolescents version) with scores that range from 6 (infrequent use of cognitive reappraisal) to 30 (frequent use of cognitive reappraisal).
Time Frame: Baseline and six month follow-up
Population: Participants who completed at least one session. By design, mothers' family members did not participate in Standard of Care intervention sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Video-based Family Therapy:Adult Mothers; Video-based Family Therapy:Adolescent Mother; Video-based Family Therapy: Family Members: Resilience Enhancement Skills Training (REST) is the family therapy intervention. Mothers and their family members participated in REST sessions. Study measures were administered to each mother and her family member, separately.
- Standard of Care:Adult Mothers; Standard of Care:Family Members: Video-based Problem-Solving individual Therapy (V-PST) is the active comparison condition. Only mothers participated in V-PST sessions. Study measures were administered to each mother and her family member, separately.
Arm/Group | Video-based Family Therapy:Adult Mothers | Video-based Family Therapy:Adolescent Mother | Video-based Family Therapy: Family Members | Standard of Care:Adult Mothers | Standard of Care:Family Members
Number analyzed (Participants) | 37 | 1 | 38 | 37 | 37
units on a scale
  Baseline | 23.5 (5.7) | 18.0 (0.0) | 28.1 (7.7) | 25.8 (5.7) | 31.6 (5.8)
  Six month follow-up: number analyzed (Participants) | 37 | 0 | 38 | 37 | 37
  Six month follow-up | 31.6 (5.8) |  | 32.5 (6.8) | 30.2 (5.4) | 34.3 (5.8)

5. Secondary Outcome: Maternal School Enrollment/Job Attainment
Description: Adapted item from ABCD study.
Time Frame: Change from baseline in maternal school enrollment/job attainment at 6 months
Population: Mothers without circumstances that prevented them from obtaining employment and enrolling in school at baseline were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based Family Therapy: Mothers | Standard of Care: Mothers
Number analyzed (Participants) | 31 | 30
Participants
  Baseline | 11 | 12
  Six month follow-up: number analyzed (Participants) | 28 | 24
  Six month follow-up | 23 | 13

ADVERSE EVENTS:
Time Frame: Nine months
Arm/Group | Video-based Family Therapy:Mothers | Video-based Family Therapy: Family Members | Standard of Care: Mothers | Standard of Care: Family Members
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 1/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT04741776/Prot_SAP_000.pdf